CLINICAL TRIAL: NCT03217500
Title: A Randomized Controlled Clinical Trial of Corneal Epithelial Autograft for Pterygium
Brief Title: Corneal Epithelial Autograft for Pterygium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chunxiao Wang (Other)
Responsible Party: Sponsor-Investigator, Chunxiao Wang, Clinical investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017KYPJ050
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Corneal epithelial autograft (Experimental): pterygium resection combined with femtosecond laser assisted corneal epithelial autograft
  Interventions: Procedure: Corneal epithelial autograft; Device: Femtosecond laser
- Limbal conjunctival autograft (Active Comparator): pterygium resection combined with diamond knife assisted limbal conjunctival autograft
  Interventions: Procedure: Limbal conjunctival autograft; Device: Diamond knife
- Simple removal (Active Comparator): Simple removal of pterygium
  Interventions: Procedure: Simple removal

INTERVENTIONS:
Procedure: Corneal epithelial autograft — After removal of the recipient's pterygium tissue, a donor epithelial tissue equal in length to the bared limbus, will be obtained from the peripheral epithelial of the same eye (corneal epithelial autograft) using femtosecond laser technology. The epithelial graft will be sutured to the recipient limbal bed, with the goal of reconstruction of palisades of Vogt. The graft will act as a barrier to regrowth of pterygium. The area of the graft will be left with the Tenon capsule exposed.
  Arms: Corneal epithelial autograft
Procedure: Limbal conjunctival autograft — After removal of the recipient's pterygium tissue, an adjustable diamond knife will be used to create a superficial circumferential incision at the corneal end of the limbal vascular arcade, equal in length to the bared limbus. This will be followed by harvesting the limbal-conjunctival flap. The limbal-conjunctival autograft will be sutured to the recipient bed, with the Tenon capsule exposed. The graft will serve as a barrier to regrowth of pterygium.
  Arms: Limbal conjunctival autograft
Procedure: Simple removal — Simple removal of the recipient's pterygium tissue, with the Tenon capsule exposed.
  Arms: Simple removal
Device: Diamond knife — A diamond knife to create a particular shaped limbal graft for transplantation
  Arms: Limbal conjunctival autograft
Device: Femtosecond laser — A commercial femtosecond laser to create a particular shaped graft for transplantation
  Arms: Corneal epithelial autograft

SUMMARY:
The purpose of the study is to explore whether femtosecond laser-assisted cornea epithelial autograft is more effective than limbal conjunctival autograft for ocular surface reconstruction after excision of pterygium.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 80 years old;
2. Primary pterygium, scheduled for elective surgical excision;
3. Pterygium encroaching from the nasal side onto the cornea, with less than 180° limbal involvement and without approaching the central visual axis (pupil area);
4. Morphologically intact palisades of Vogt in a given limbal region;
5. Absence of any one of the following structures in the limbal region underneath the pterygium: (1) epithelial basal cells with dark cytoplasm and reflective cell borders; (2) at least two prominent palisade ridge structures; (3) at least one circular and/or oval-shaped focal stromal projection;
6. Informed consent signed by patient or legal guardian; Having the ability to comply with study assessments for the full duration of the study.

Exclusion Criteria:

1. Limbal stem cell deficiency by ocular surface disorders other than pterygium;
2. Inability to determine whether the palisades of Vogt underneath the pterygium is absent or not using in vivo confocal microscopy;
3. High myopia with a spherical equivalent of -15.0 D or less;
4. Corneal or ocular surface infection within 30 days prior to study entry;
5. Ocular surface malignancy;
6. Uncontrolled diabetes with most recent Hemoglobin A1c greater than 8.5%;
7. Renal failure with creatinine clearance< 25ml/min;
8. Alanine aminotransferase > 40IU/L, or aspartate aminotransferase > 40IU/L;
9. Platelet levels < 150,000 or > 450,000 per microliter;
10. Hemoglobin < 12.0 g/dL (male) or < 11.0 g/dL (female);
11. Prothrombin time > 16s and activated partial thrombin time > 35s in patients not accepting anticoagulant therapy; An international normalized ratio greater than 3 in patients accepting anticoagulant therapy;
12. Pregnancy (positive test) or lactation;
13. Participation in another simultaneous medical investigation or clinical trial;
14. Severe cicatricial eye disease;
15. Ocular comorbidities that affect the prognosis of transplantation, such as advanced glaucoma or retinal diseases;
16. Severe dry eye disease as determined by Schirmer's test < 2mm at least in one eye;
17. Any medical or social condition that in the judgement of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent;
18. Signs of current infection, including fever and treatment with antibiotics;
19. Active immunological diseases;
20. History of allo-limbal transplantation, penetrating keratoplasty or anti-glaucoma filtering surgeries.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Restoration of corneal surface | 1 year
  Restoration of a completely epithelized, stable, and avascular corneal surface

SECONDARY OUTCOMES:
Recurrence of pterygium | 1 year
  To observe recurrence of pterygium using slit-lamp microscopy
Reconstruction of palisades of Vogt | 1 year
  To observe the reconstruction of palisades of Vogt using in vivo confocal microscopy.
Best corrected visual acuity | 1 year
  To assess changes of best corrected visual acuity using ETDRS chart
Corneal power and astigmatism | 1 year
  To assess changes of corneal power and astigmatism using autorefractor keratometer
Corneal haze measurement | 1 year
  To observe the scatter of corneal haze using in vivo confocal microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Ting Huang, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China